CLINICAL TRIAL: NCT00493077
Title: A Swedish Multi-Centre, Prospective, Open Label Study: Safety of Avonex Treatment in Multiple Sclerosis Patients Who Are NAB Positive on Previous s.c Interferon Beta Therapy
Brief Title: Safety of Avonex Treatment in Multiple Sclerosis Patients With Neutralizing Antibodies to Interferon Beta Therapy
Acronym: SAFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: biogen Idec MD, Biogen Idec
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFE
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Neutralizing antibodies; Safety; Low immunogenicity; interferon; interferon-beta-1a
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: low immunogenic interferon-beta-1a

INTERVENTIONS:
Drug: low immunogenic interferon-beta-1a — dosage and frequency as per Biogen Idec protocol
  Other Names: Avonex

SUMMARY:
This study is to find out the safety and effectiveness of Avonex (interferon-beta-1a) Therapy in patients who have developed neutralizing antibodies during previous interferon-beta treatment

DETAILED DESCRIPTION:
This is a multi-centre, prospective, open label, non-comparative phase IV trial. Eligible patients will receive treatment with IFN-beta-1a AVONEX® 30 mcg i.m. once weekly for 12 months.The patients will be examined clinically and NAb titres will be performed at screening and after 12 months. Adverse event source verification will be performed during the documentation period.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting MS according to Poser criteria(CDMS or LSDMS)30 or MS according to McDonald criteria
* Disability equivalent to an EDSS of 6.0 or less at screening
* Neutralizing antibody titre > 20 and <500 in two consecutive NAb tests. One must be from before screening
* previous treatment with either subcutaneous administered interferon-b-1b (Betaferon®) or interferon-b-1a (Rebif TM) prior to enrolment
* A priori has been decided to be treated with AVONEX

Exclusion Criteria:

* Is NAb positive on AVONEX
* History of major depression
* Cardiac insufficiency, cardiomyopathy, significant cardiac dysrhythmia, unstable or advanced ischemic heart disease (NYHA III or IV), or significant hypertension (BP > 180/110 mmHg)
* Renal insufficiency defined as serum creatinine > 1.5 times the upper normal reference limit
* Any systemic disease that can influence the patient's safety and compliance, or the evaluation of the disability
* Women who are pregnant, breast-feeding or have the possibility for pregnancy during the trial. To avoid pregnancy, women have to be postmenopausal, surgical sterile, sexually inactive or practice reliable contraceptives

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2004-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
neutralizing antibody levels will be followed | 12 months

SECONDARY OUTCOMES:
Proportion of patients with NAb positive titre > 20. | 12 months
Relative change from baseline (screening) of NAb titre | 12 months
Change in the annualised relapse rate and number of relapse-free (total and documented relapses) patients | 12 months and as needed for relapses
The percentage of patients with a loss of disability of 1.0 (or more) score on the EDSS. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Principal Investigator — neurologyclinicaltrials@biogenidec.com
Locations (5):
- Sweden (5):
  - Research Site, Gothenburg
  - Coordinating Research Site, Huddinge
  - Research Site, Jönköping
  - Research Site, Karlstad
  - Research Site, Stockholm